CLINICAL TRIAL: NCT06603792
Title: Neurofeedback for the Management of Neuropathic Pain in People with Diabetes
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: European Foundation for the Study of Diabetes (Other); Region of Southern Denmark (Other); Vissing fonden (Unknown); Steno Diabetes Center Odense (Other); Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Francois Pouwer, Professor, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11.719
Record Dates: First submitted 2024-08-29; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-05

CONDITIONS: Neuropathy, Painful Diabetic
Keywords: Neurofeedback; diabetic neuropathy; painful diabetic neuropathy; RCT; EEG-neurofeedback
MeSH Terms: conditions — Diabetic Neuropathies

STUDY DESIGN:
Intervention Model Description: The project will investigate two randomized groups: a 'true' EEG-NF-group and 'sham' EEG-NF-group.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Real EEG-neurofeedback (Experimental): the NF intervention group will receive feedback based on the genuine real-time EEG activity
  Interventions: Behavioral: EEG-neurofeedback
- Sham EEG-neurofeedback (Sham Comparator): The sham-group will receive another participant's EEG-training protocol as a prerecorded signal. The feedback signal will consist of 15-25 rewards per minute. Meanwhile, the threshold for the sham group remains fixed, ensuring a consistent 70% positive feedback rate.
  Interventions: Behavioral: EEG-neurofeedback

INTERVENTIONS:
Behavioral: EEG-neurofeedback — Traditional neurofeedback uses one or two electrodes to modulate activity within a specific frequency band. Standardized Weighted Low Resolution Electromagnetic Tomography (swLORETA) analyzes the 3D distribution of intracortical brain electrical activity based on surface EEG recordings, enabling real-time brainwave imaging with a spatial resolution under one cubic centimeter. This divides the brain into over 12,000 voxels, offering localization similar to fMRI while maintaining EEG's faster temporal resolution. Source-localized NF can target specific, deeper brain regions, multiple Brodmann areas simultaneously, and provide feedback on connectivity between neural sources, enabling the training of specific neural networks. swLORETA metrics are compared to a normative database of neurotypical brains to produce z-scores for each area and metric. We will use the NeuroGuide normative database, FDA-approved and validated in peer-reviewed studies, widely used in clinical NF.

SUMMARY:
We will conduct a high-quality, blinded, randomized controlled trial (RCT) to rigorously test the effectiveness of EEG-based NF in patients with diabetes-related neuropathic pain in: 1) reducing pain intensity and pain affect, and 2) improving daily functioning and QoL.

DETAILED DESCRIPTION:
20%-40% of people with diabetes develop diabetic polyneuropathy (DPN), which often manifests as a painful complication, strongly reducing quality of life. Current standard pharmacological treatments for neuropathic pain are often ineffective and have considerable side effects. Therefore, there is an urgent need for better treatment options. The way in which the brain interprets signals from the periphery can be modified through learning certain techniques, which can enable patients to modify signals related to painful DPN and consequently experience pain alleviation. Neurofeedback (NF) is a promising neuromodulatory therapy in which individuals receive real-time feedback about their brain's neurophysiological signals, thus increasing the volitional control of brain activity, reducing the experience of pain. Neurofeedback uses scalp EEG electrodes attached to a computer screen, which give real-time feedback to the individual. NF may offer symptom alleviation by teaching patients to regulate relevant activity patterns by themselves. By rewarding the person whenever the neural activity changes in a desired direction, the activity can be modulated. NF has not yet been investigated in an RCT in people with painful DPN. This proposed Danish-Brazilian project is the first triple blind RCT rigorously testing an EEG-NF intervention for neuropathic pain (NP) in diabetes. The treatment will be conducted over 10 sessions in two randomized groups: a real EEG-NF group and a sham (placebo) EEG-NF group. Brazilian participants will also undergo (functional) magnetic resonance imaging (fMRI) scanning to investigate how the NF-treatment targets and alters neural mechanisms. If found effective, the low-cost EEG-NF can be made available and implemented at large scale for people with diabetes and painful neuropathy, and will be in reach for low- to middle-income countries.

ELIGIBILITY:
Inclusion Criteria:

Age ≥18 and ≤82 years

* Diagnosed with 1) type 1 diabetes (for at least 5 years) or 2) type 2 diabetes
* The Toronto consensus criteria will be used for a case definition of DPN where patients have to have at least probable DPN (31). Diagnosis of DPN is confirmed with abnormal DPN Check. Painful DPN will be defined using the grading system for neuropathic pain (50) and will be in line with IASP's definition of neuropathic pain, i.e., "pain caused by a lesion or disease of the somatosensory system" (The Toronto consensus criteria).
* TCNS score > 5
* Eligible patients with painful DPN must have a pain intensity of at least 4 on an 11-point numerical rating scale (NRS, 0-10) for at least 3 months on at least semi-daily basis and no severe pain other than pain due to neuropathy (the pain intensity will be based on the pain the patients experience while on current pain treatment, if any).
* Stable pain medication for > 1 month prior to inclusion. Exclusion criteria

Exclusion Criteria:

* Concomitant neurological (neurodegenerative disorders, migraine, epilepsy, stroke, tumor) or clinically significant psychiatric illness
* Neuropathy or neuropathic pain due to other causes than diabetes (vitamin B12 deficiency, prior treatment with neurotoxic chemotherapy, chronic alcohol abuse, spinal stenosis, etc.)
* Change in current pain treatment during treatment (paracetamol is allowed as rescue medicine)
* Prior or current excessive alcohol use (>14 or >21 units/week for women and men, respectively) or illegal substance abuse
* Positive urine hCG test result indicating pregnancy
* Morphine use >20mg/day
* Blindness or severely impaired vision
* The investigator finds the patient unfit for the study (e.g. due to use of alcohol or drugs, mental incapacity, unwillingness, or language barrier precluding adequate understanding or cooperation or presence of any condition that in the investigators' opinion may lead to poor adherence to study protocol).

Ages: 18 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Pain intensity and affect | Before and after the intervention (approx. 8 weeks)
  Change in self-reported pain intensity and pain affect (an average over a daily measurement in a 7-day pain diary using a numeric rating scale (NRS) from 0-10)

SECONDARY OUTCOMES:
Neuropathic pain severity | Before and after the intervention (approx. 8 weeks) and at 4 months follow-up (approx. a half year from start until four months follow up)
  Differences in neuropathic pain severity as measured by PROMIS. Both individually and between groups
Neuropathic pain severity | Before and after the intervention (approx. 8 weeks) and at 4 months follow-up (approx. a half year from start until four months follow up)
  Differences in neuropathic pain severity as measured by the DN4. Both individually and between groups
Neuropathic pain severity | Before and after the intervention (approx. 8 weeks) and at 4 months follow-up (approx. a half year from start until four months follow up)
  Differences in neuropathic pain severity as measured by the Neuropathic pain severity as measured by the Neuropathic Pain Scale (NPS). Both individually and between groups
Disability | Before and after intervention (approx. 8 weeks). Between groups after intervention (approx. 8 weeks) and at 4 months follow-up (approx. a half year after baseline)
  Differences in disability as measured by the Brief Pain Inventory (BPI) (short form) and on the full BPI.
Sleep quality | 7 day diary before baseline and after intervention (approx. 8 weeks)
  Daily sleep interference scale
z-score normalization | Before and after the intervention (approx. 8 weeks)
  Normalization of the z-score of the targeted neural networks described in the training protocol for the NF-treatment.
Loreta z-score responders versus non-responders | Before and after the intervention (approx. 8 weeks)
  Investigate Loreta z-score responders versus non-responders. Responders will be a subgroup of participants who showed any amount of decrease from baseline to last visit in the total number of significant z-scores within the targeted networks. Responders, whose z-scores move toward neurotypical levels (i.e., toward z = 0) will be compared to non-responders whose z-scores will not move in this expected direction.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Southern Denmark, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No